CLINICAL TRIAL: NCT05655663
Title: Evaluation of Vascular Toxicity of Immune Checkpoint Inhibitors (Nivolumab, Pembrolizumab, Atezolizumab) in Patients Head and Neck or Lung Cancer
Brief Title: Evaluation of Vascular Toxicity of Immune Checkpoint Inhibitors in Patients Head and Neck or Lung Cancer
Acronym: IMMUNOVASC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB19.02
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Cancer; Lung Cancer
Keywords: immune checkpoint inhibitor; head and neck cancer; lung cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICI (Experimental): Patients under ICI treatment for their cancer will have vascular investigation and biological assessment
  Interventions: Other: Vascular investigation

INTERVENTIONS:
Other: Vascular investigation — Measure of of carotid stiffness

SUMMARY:
Since the introduction of immune checkpoint ihibitors (ICIs) in cancer treatment, numerous studies have investigated different patient profiles to identify those who benefit from this class of drugs. Currently, hundreds of studies are being conducted with the aim of increasing the benefit of these therapies by combining ICIs with other treatments: immunomodulators, cytotoxics, targeted therapies, including cancer vaccines, which are peptides or RNA injected to trigger or increase a specific immune response against the tumor. Other approaches exist, such as oncology-specific "basket" studies, to focus on a genetic mutation independently of tumor location and determine whether a drug could treat the same genetic mutation found in several different locations. To date, ICIs are part of standard management in the US for patients with several diseases: advanced melanoma, NSCLC, Merkel cell carcinoma, head and neck squamous cell carcinoma, urothelial and renal cell carcinoma, cancers characterized by microsatellite instability, refractory Hodgkin's lymphoma, hepatocellular carcinoma, gastric cancer. In addition, trials are underway to investigate the benefit of ICIs in other locations.

Thus, taking into account the growing importance of ICIs in the oncological therapeutic strategy and the large number of patients treated, a better understanding of the vascular impact of these drugs is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Patient over 18 years of age
* Patient with lung or head and neck cancer who should be treated with ICI as a single agent according to the market indications, decision taken during a multidisciplinary consultation meeting
* WHO 0 or 1
* Patient affiliated to or benefiting from a social protection scheme.

Exclusion Criteria:

* Indication for combined anti-PD-1 and chemotherapy (for patients with lung cancer)
* History of radiotherapy treatment
* History of chemotherapy or targeted therapy within the last 3 weeks
* Bilateral vascular carotid murmur
* Absence of sinus rhythm
* Presence of a pacemaker with permanent electrical stimulation
* Absence of peripheral carotid and/or femoral pulses on both sides
* Contraindication to the prescription of an ICI
* Patient deprived of liberty by an administrative or judicial decision or patient placed under court protection, guardianship or curatorship
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Increasing of aortic arterial stiffness | 42 days
  Difference of aortic arterial stiffness between 42 days after inclusion and inclusion

SECONDARY OUTCOMES:
Overall survival | one year
  Time between death and inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Olympios, MD, Principal Investigator — Centre Henri Becquerel
Locations (2):
- France (2):
  - Centre Henri Becquerel, Rouen
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No